CLINICAL TRIAL: NCT05703035
Title: The Effects of Waiting 1 Minute During Stapling During Laparoscopic Sleeve Gastrectomy on
Brief Title: Waiting for Stapler Firing in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medeni Şermet (Other)
Responsible Party: Sponsor-Investigator, Medeni Şermet, specialist general surgery, Goztepe Prof Dr Suleyman Yalcın City Hospital
Organization: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021/0530
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Staple Misfire

STUDY DESIGN:
Intervention Model Description: Two equal groups with equal comorbid conditions will be compared
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Computer-assisted 4-block-based randomization via random.org
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- waiting group during staple firing (Active Comparator): In this group, the amount of bleeding, bleeding points, postoperative drain amount and laboratory values will be monitored during the operation.
  Interventions: Procedure: standby while firing staple
- staple firing group without waiting for a certain time (Active Comparator): In this group, no further intervention will be made, and the same treatment will be given as the 1st group and comparison will be made.
  Interventions: Procedure: standby while firing staple

INTERVENTIONS:
Procedure: standby while firing staple — VOLUNTEER PATIENTS WHO ACCEPT THE SURGERY WILL HAVE TISSUE CLOSURE AND CUTTING WITH STAPLER IN AVERAGE 30 MINUTES DURING THE SURGERY AND THE PATIENT WILL BE FOLLOWED FOR 30 DAYS.

SUMMARY:
Complications will be evaluated by waiting 30 seconds after firing 30 seconds during stapler compression while performing sleeve gastrectomy.

DETAILED DESCRIPTION:
Those with a BMI between 35.0 and 39.90 and those with an obesity-related comorbidity, and all morbid obesity patients with a BMI of 40.0 and above, were previously adequate for at least 6 (six) months with non-surgical (diet, medication, exercise, etc.) methods. Patients with morbid obesity who could not lose weight and who were unsuccessful will be included in the study by signing an informed consent form for the operation and study, after being evaluated by the "obesity council" consisting of endocrinology, psychiatry, anesthesiology, dietitian and general surgery, and approved for bariatric surgery. Waiting will be made for patients whose patient file number has an odd number in the last digit, and no waiting will be made for patients whose last digit is an even number. At the time of the operation, the patients will be put on thromboembolic stockings and the reverse trendelenburg position will be given and the operation will be started with the laparoscopic method. After the stomach is mobilized from the adjacent organs and structures, the 38F gastric tube will be advanced to the stomach, the tissue will be closed with a 60 mm laparoscopic stapler, waited for 30 seconds, and then ignition will be performed. After the stapler is fired, a waiting period of 30 seconds will be waited and it will be removed from the tissue. In this first case, whether there is bleeding or not, at how many points, whether additional intervention is required or not will be recorded. At the end of the operation, the gastric tube will be withdrawn, and the stomach will be filled with 120 cc saline colored with methylene blue to check if there is any leakage. If there is no leakage, a gastric drainage drain will be placed and the operation will be completed. Postoperative 24 - 48 . After discharge, the patient will be called for routine control on the 1st week, 15th day and 30th day after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Among the patients between the ages of 18-65 who will undergo morbid obesity operation;

  1. Body mass index (BMI): 35.0-39.9 and those with at least one obesity-related comorbidity
  2. Patients with BMI: 40.0-49.9

Exclusion Criteria:

* a-Applicants for revision surgery, b- Patients with a history of thromboembolism, c- Patients with known coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
to measure that waiting a certain time before and after firing the stapler can reduce complications. | the period from the 1st day to the 1st month postoperatively will be taken as a basis.
  There will be a waiting period of 30 seconds during stapler compression and 30 seconds after ignition. Thus, complications such as postoperative bleeding and leakage can be reduced.

CONTACTS AND LOCATIONS:
Overall Officials: medeni sermet, 1, Study Director — goztepe prof. dr. suleyman yacin city hospital
Locations (1):
- Medeni Sermet, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sermet M. Compression pre-stapler firing and post-ignition wait during sleeve gastrectomy: a prospective randomized trial. Sao Paulo Med J. 2023 Dec 15;142(3):e2023163. doi: 10.1590/1516-3180.2023.0163.140823. eCollection 2023. PMID 38126605